CLINICAL TRIAL: NCT02503943
Title: What is the Effects of Incretin on the Blood Pressure and Lipid in Overweight or Obese Diabetes Patients With Masked Hypertension: Liraglutide Plus Mitiglinide Comparing Metformin Plus Mitiglinide or Mitiglinide Alone（BLOOD STUDY）
Brief Title: Effects of Incretin on the Blood Pressure and Lipid in Patients With Overweight or Obese Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Third Affiliated Hospital of Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yinxing Ni, Medical Doctor, Third Affiliated Hospital of Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLOOD
Record Dates: First submitted 2015-05-13; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes; Overweight; Obesity; Masked Hypertension
Keywords: GLP-1; Masked hypertension; Lipid metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Masked Hypertension | interventions — Liraglutide; mitiglinide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- "Liraglutide" and "Mitiglinide" (Experimental): "Liraglutide"(1.2mg/d) and "Mitiglinide"(50mg, 3/d)
  Interventions: Drug: "Liraglutide" and "Mitiglinide"
- "Metformin" and "Mitiglinide" (Active Comparator): "Metformin"(500mg, 3/d) and "Mitiglinide"(50mg, 3/d)
  Interventions: Drug: "Metformin" and "Mitiglinide"
- "Mitiglinide" (Active Comparator): "Mitiglinide"(50mg, 3/d)
  Interventions: Drug: "Mitiglinide"

INTERVENTIONS:
Drug: "Liraglutide" and "Mitiglinide" — "Liraglutide"(1.2mg/d) and "Mitiglinide" (50mg, 3/d)
  Arms: "Liraglutide" and "Mitiglinide"
Drug: "Metformin" and "Mitiglinide" — "Metformin"(500mg, 3/d) and "Mitiglinide"(50mg, 3/d)
  Arms: "Metformin" and "Mitiglinide"
Drug: "Mitiglinide" — "Mitiglinide" (50mg, 3/d)
  Arms: "Mitiglinide"

SUMMARY:
Obesity is one of the characteristics of type 2 diabetes mellitus. Most of the obese diabetes patients are combined with dyslipidemia or hypertension. The clustering of diabetes, obesity, hypertension and dyslipidemia increases the risk of cardiovascular events for patients. GLP-1 (glucagon like peptide-1) is a kind of incretin discovered in recent years. It was reported that beside its hypoglycemic and losing weight effects, activator of GLP-1 receptor could decrease blood pressure and improve lipid metabolism. Therefore, activation of GLP-1 receptor may become a new comprehensive treatment strategies for improving glucose and lipid metabolism, blood pressure level and cardiovascular complication. But, it is lack of evidence-based medicine proof on the relationship between GLP-1 and blood pressure or serum lipid. So, investigators designed a prospective, randomized, open-label, active control study, and try to evaluate the effects of activator of GLP-1 receptor (liraglutide) on lowering blood pressure, improving vascular function and lipid metabolism in overweight or obese type 2 diabetic patients with masked hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age between 35-60 years old
2. Type 2 diabetes
3. 24kg/m²≤BMI≤32kg/m², or WC≥90cm for male and WC≥85cm for female
4. Grade 1 hypertension or masked hypertension diagnosed via 24-h ambulatory blood pressure monitoring (daytime blood pressure load 50%≥135/85 mmHg, night time blood pressure load 50%≥125/75 mmHg or 24h blood pressure load 50%≥130/80 mmHg）

Exclusion Criteria:

1. Type 2 diabetes with serious complications, such as diabetic neuropathy, diabetic retinopathy, stage IV diabetic nephropathy, or acute diabetic complications.
2. Type 1 diabetes.
3. Diagnosed moderate to severe sleep apnea syndrome(SAS).
4. Grade 2 or Grade 3 hypertension.
5. Triglyceride≥5.65mmol/L
6. History of cardio-cerebral vascular events such as congestive heart failure, myocardial infarction or stroke within 3 months.
7. Hypohepatia (AST or AST is twice higher than the upper limit) or history of hepatitis or cirrhosis, hepatic encephalopathy.
8. Renal insufficiency ( serum creatinine is 1.5 times higher than the upper limit) or history of dialysis and nephritic syndrome.
9. Chronic obstructive pulmonary disease (COPD), chronic respiratory failure or hyoxemia.
10. Acute infections, tumor, severe arrhythmia, mental disorders, alcohol or medicine addiction.
11. Fertile woman without contraceptives.
12. Any surgical or medical conditions that significantly influence absorption, distribution, metabolism or excretion of the intervention drugs.
13. Allergic to or have contraindication to the intervention drugs.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure change | Baseline,4 weeks,8 weeks,12 weeks,16 weeks,20 weeks,up to 24 weeks
Lipid profile (triglyceride, total cholesterol, LDL-c; HDL-c; mmol/L) change | Baseline,4 weeks,8 weeks,12 weeks,16 weeks,20 weeks,up to 24 weeks

SECONDARY OUTCOMES:
24-hours mean blood pressure; incidence of clinical hypertension; Blood pressure variability, Heart rate variability. | Baseline，12 weeks,up to 24 weeks
Hemodynamics parameters, including pulse wave velocity(PWV) | Baseline,4 weeks,8 weeks,12 weeks,16 weeks,20 weeks,up to 24 weeks
24-hours urine sodium and microalbumin | Baseline,4 weeks,8 weeks,12 weeks,16 weeks,20 weeks,up to 24 weeks
Carotid intima-media thickness(IMT,mm) | Baseline，12 weeks,up to 24 weeks
Obesity parameters, including waist circumference (WC,cm) and body mass index(BMI, kg/m2) | Baseline,4 weeks,8 weeks,12 weeks,16 weeks,20 weeks,up to 24 weeks
Insulin resistance assessed by fasting serum insulin and HOMA-IR, and control rate of diabetes. | Baseline,4 weeks,8 weeks,12 weeks,16 weeks,20 weeks,up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Zhu, MD, PHD, Study Chair — The third hospital affiliated to the Third Military Medical University. China